CLINICAL TRIAL: NCT04501926
Title: Genomics and Metagenomics of Asthma Severity
Acronym: GEMAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maria Pino-Yanes (Other)
Collaborators: University of La Laguna (Other); Ministry of Science and Innovation, Spain (Other Government); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); University Hospital of the Nuestra Señora de Candelaria (Other); Hospital Universitario de Canarias (Other); Hospital General de La Palma (Unknown); Hospital Donostia (Other); Hospital Doctor Jose Molina Orosa (Unknown)
Responsible Party: Sponsor-Investigator, Maria Pino-Yanes, Ramon y Cajal Fellow and Lecturer, University of La Laguna
Organization: University of La Laguna (Other)
Other Study IDs: PI-29/17
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Asthma; Asthma Attack
Keywords: Genome-Wide Association Study; Microbiome, Human; Asthma; Epigenomics; Transcriptomics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples are drown in EDTA tubes and PAXGene tubes for human DNA and RNA extraction, respectively. For the human microbiome study, saliva samples and nasal and pharyngeal swaps are collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Asthma patients who did not report asthma exacerbations in the 12 months prior recruitment, defined by one of the following events because of asthma: oral corticosteroids use, emergency room visits, and/or hospitalizations.
- Cases: Asthma patients that reported asthma exacerbations in the 12 months prior recruitment, defined by one of the following events because of asthma: oral corticosteroids use, emergency room visits, and/or hospitalizations.

SUMMARY:
The Genomics and Metagenomics of Asthma Severity (GEMAS) study aims to assess the role of genomics, the microbiome, and the interaction between them in the development of asthma exacerbations in European patients with asthma.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease of the airways characterized by reversible airflow obstruction and a bronchial hyperreactivity in response to a variety of stimuli. In most patients, the onset of asthma symptoms may be controlled. However, many of them may manifest asthma attacks or crises of breathing called exacerbations, which occur with breathing problems, wheezing, coughing or tightness of chest, and may threaten their life. Such exacerbations are caused by a combination of environmental and genetic factors. However, since studies so far have been limited, a reduced number of genes associated with the predisposition to these complications have been identified. In addition, some studies have used next-generation DNA sequencing techniques to characterize the microbiome (i.e., microbial community) of the airways, finding changes related to asthma. The main hypothesis of the Genomics and Metagenomics of Asthma Severity (GEMAS) study is that exacerbations of asthma are caused by a combination of the intrinsic genetic factors of the individual, changes in the respiratory microbiome and the interaction between both factors. The objectives of this project are: 1) to identify genetic variants that are associated with asthma exacerbations; 2) to examine the changes occurring in the microbial communities of the oral cavity and respiratory tract in individuals with exacerbations; 3) to analyze the association of the host genetic variants and the microbiome changes related to exacerbations.

A total of 300 Spanish subjects with asthma with and without a history of asthma exacerbations in the past 12 months will be recruited. Saliva, nasal and pharyngeal samples will be collected to study the oral cavity and the upper respiratory tract microbiome through next-generation sequencing technologies. Sequencing of the 16S ribosomal RNA (16S rRNA) gene will allow to characterize the bacterial diversity and abundance, as well as to infer the functionality of the microbiome in each sample. These parameters will be used to establish correlations between the microbiome and the presence of asthma exacerbations. Finally, the association between the genetic variation associated with exacerbations in genomic studies and the measurements of abundance, diversity and functions related to exacerbations will be jointly examined.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged older or equal than 8 years and younger or equal than 85 years
* Physician diagnosis of asthma according to the Global Initiative for Asthma (GINA) guidelines
* Treated on GINA step 1-5

Exclusion Criteria:

* One or more grandparents of non-European origin
* Pregnancy
* Coexistence of other chronic pulmonary disorders including cystic fibrosis, chronic obstructive pulmonary disease (emphysema or chronic bronchitis), or congenital disorders of the lungs or airways
* Known family relatedness (first or second degree) with another participant already included in the study

Ages: 8 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are recruited from the allergy and/or pulmonary medicine units from hospitals located in the Canary Islands, Spain (Hospital Universitario de Canarias, Hospital Universitario Nuestra Señora de Candelaria, Hospital General de La Palma, and Hospital Doctor Jose Molina Orosa), and in the division of pediatric respiratory medicine of Hospital Universitario Donostia in the Basque Country, Spain.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Severe asthma exacerbations | 1 year
  Defined by one of the following events because of asthma during the past year, the past 6 months, and the past week: oral corticosteroids use, emergency room visit, and/or hospitalizations

SECONDARY OUTCOMES:
Asthma control | 1 week
  Asthma control questionnaire (ACQ) score
Asthma severity | 1 year
  Category of severity defined by treatment step according to GINA 2020 at recruitment
Lung function measurement: forced expiratory volume in the first second (FEV1) | 3 months
  Baseline and post-bronchodilator measurements of the forced expiratory volume in the first second (FEV1) measured in liters
Lung function measurement: forced vital capacity (FVC) | 3 months
  Baseline and post-bronchodilator measurements of the forced vital capacity (FVC) measured in liters
Lung function measurement: FEV1/FVC ratio | 3 months
  The ratio of FEV1/FVC measurements
Atopy testing | 1 year
  Atopy status evaluated by skin prick tests and/or specific immunoglobulin E (IgE) levels assessing the most common aeroallergens of each recruiting center

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - University of La Laguna, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Doctor Jose Molina Orosa, Arrecife
  - Hospital General de La Palma, Breña Alta
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife

IPD SHARING:
Plan to Share IPD: No